CLINICAL TRIAL: NCT06744595
Title: Evaluation of Genetic Testing for Patients With Known Family History of Pancreatic Cancer: A Pilot Study
Brief Title: Personalized Education and Genetic Counseling to Increase Genetic Testing in Patients With a Known Family History of Pancreatic Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-006906; NCI-2024-10177 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-006906 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Specimen Handling; Early Intervention, Educational; Educational Status; Methods; Genetic Counseling; Genetic Testing; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Health services research (EPIC message, genetic counseling) (Experimental): Patients receive a personalized message through EPIC with education on the NCCN guidelines for genetic counseling and an offer for SOC genetic counseling. Patients then receive pre-genetic test counseling on study. Patients may then optionally undergo SOC genetic testing and collection of blood or saliva samples as well as receive post-genetic test counseling on study.
  Interventions: Procedure: Biospecimen Collection; Other: Educational Intervention; Other: Electronic Health Record Review; Other: Genetic Counseling; Genetic: Genetic Testing for Cancer Risk; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood or salvia samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Educational Intervention — Receive personalized EPIC message
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Electronic Health Record Review — Ancillary studies
Other: Genetic Counseling — Receive pre-genetic test counseling
Other: Genetic Counseling — Receive post-genetic test counseling
Genetic: Genetic Testing for Cancer Risk — Undergo SOC genetic testing
  Other Names: Cancer Risk Assessment with Genetic Testing and Counseling
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial studies whether personalized education and genetic counseling increases genetic testing in patients with a known family history of pancreatic cancer. Approximately 10% of pancreatic cancer cases are genetically linked and therefore, if a gene is found that could put a patient at risk, it could guide the patient to obtain more frequent screening for pancreatic cancer and possibly detect it earlier when it is more treatable. The current National Comprehensive Cancer Network (NCCN) guidelines suggest patients with a first-degree relative (parent, sibling, child) with pancreatic cancer be referred for a genetics consultation to discuss genetic testing if the affected family member cannot be tested. Personalized education is based on the patient's family history of pancreatic cancer and offers information regarding the current NCCN guidelines. This may be an effective method to increase patients' understanding of their pancreatic cancer risk and the NCCN guidelines. Genetic counseling is provided by an expert in hereditary disorders. The patient's family and personal medical history may be discussed, and counseling may lead to genetic testing. Personalized education and genetic counseling may increase genetic testing in patients with a known family history of pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Perform Housing-Based Socioeconomic Status (HOUSES) index analysis on 500 patients with a first-degree relative diagnosed with pancreatic cancer to see if there is a correlation with the National Comprehensive Cancer Network (NCCN) criteria.

II. Offer 40 patients who did not have appropriate NCCN intervention the opportunity to have a genetic consultation (to consider genetic testing).

III. Survey patients on their knowledge and experiences of genetic testing based on family history and their decision-making when offered genetic counseling and testing.

OUTLINE:

Patients receive a personalized message through the Mayo portal (EPIC) with education on the NCCN guidelines for genetic counseling and an offer for standard of care (SOC) genetic counseling. Patients then receive pre-genetic test counseling on study. Patients may then optionally undergo SOC genetic testing and collection of blood or saliva samples as well as receive post-genetic test counseling on study.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years of age
* First-degree relative with pancreatic cancer listed in the EPIC family history tool
* Active patient at Mayo Clinic Florida (MCF) (visits within 1/1/2023-12/31/2023 to Family Medicine and/or Gastroenterology and Hepatology)

Exclusion Criteria:

* Patients not meeting the inclusion criteria as defined above
* Patients with an active or past history of pancreatic cancer
* Patients who are pregnant or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Demographic factors affecting likelihood of patients meeting National Comprehensive Cancer Network (NCCN) guidelines | Up to 75 days
  Will determine whether demographic factors, including socioeconomic status, affect the likelihood of a patient meeting NCCN guidelines regarding genetic counseling for those with a family history of pancreatic cancer.

SECONDARY OUTCOMES:
Number of patients meeting NCCN guidelines | Up to 75 days
  Will determine if portal message communication can improve the number of patients who meet NCCN guidelines at Mayo Clinic in Florida and understand their experiences.

CONTACTS AND LOCATIONS:
Overall Officials: Adrianna D. Clapp, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials